CLINICAL TRIAL: NCT01525901
Title: A Double-Blind Placebo-Controlled Crossover Trial of Insulin-Like Growth Factor-1 (IGF-1) in Children and Adolescents With 22q13 Deletion Syndrome(Phelan-McDermid Syndrome)
Brief Title: Clinical Trial in 22q13 Deletion Syndrome(Phelan-McDermid Syndrome)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alexander Kolevzon, Principal Investigator, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 12-0929; IF# 1358648; 1R34MH100276-01 (NIH); GCO 11-1555 (Other: Icahn School of Medicine at Mount Sinai); R34MH100276 (NIH)
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Results first posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-04

CONDITIONS: 22q13 Deletion Syndrome; Phelan-McDermid Syndrome
Keywords: SHANK3; IGF-1; Autism
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome; Autistic Disorder | interventions — Insulin-Like Growth Factor I; mecasermin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin-Like Growth Factor-1 (IGF-1) (Experimental): Injection
  Interventions: Drug: Insulin-Like Growth Factor-1 (IGF-1)
- Normal saline (Placebo Comparator): Injection
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Insulin-Like Growth Factor-1 (IGF-1) — IGF-1 and placebo will each be administered for 3 months with a four-week washout period in between. IGF-1 will be administered for 3 months subcutaneously.
  Other Names: Mecasermin; Increlex
  Arms: Insulin-Like Growth Factor-1 (IGF-1)
Drug: Normal saline — Saline solution will be administered for three months subcutaneously.
  Other Names: Placebo
  Arms: Normal saline

SUMMARY:
The purpose of this study is to pilot the use of Insulin-Like Growth Factor-1 (IGF-1) treatment in 22q13 Deletion Syndrome (Phelan-McDermid Syndrome) caused by SHANK3 gene deficiency in order to evaluate safety, tolerability, and efficacy. IGF-1 is an injection under the skin that contains human IGF-1. IGF-1 is approved by the FDA under the brand name Increlex for the treatment of children with short stature due to primary IGF-1 deficiency. It is being used off-label in the current study and is not FDA approved, nor has it yet been studied in humans for the treatment of SHANK3 deficiency.

DETAILED DESCRIPTION:
Overall, there will be 1-3 screening visits, a baseline visit where study drug will first be administered, and then 10 follow-up visits. Follow-up visits will occur at week 2, week 4, week 8, and week 12 in each treatment phase (IGF-1 or placebo), and then again 4 weeks after study completion, Parents/guardians will be asked to administer the IGF-1/ placebo by injection at home and will also be responsible for monitoring glucose levels in the child. Parents/guardians will be trained in these methods, and will have scheduled phone calls and appointments where the dose and tolerability will be discussed.

Assessments include the following:

* Physical and neurological examination
* Medical and psychiatric history
* X-ray of long bone (e.g., hand) to ensure your child's growth plates are not closed
* Electrocardiography
* Echocardiography
* Pregnancy test if applicable
* Lab safety measures (through blood draw)
* Autism Diagnostic Interview (ADI)
* Autism Diagnostic Observation Schedule (ADOS)
* The Mullen Scales of Early Learning or the Leiter International Performance Scale-Revised
* Vineland Adaptive Behavior Scale (VABS)
* Clinical Global Impressions (CGI) Rating Scales
* The Repetitive Behaviors Scale (RBS)
* Aberrant Behavior Checklist (ABC)
* The Caregiver Strain Questionnaire (CSI)
* Language Environment Analysis (LENA)
* The Macarthur-Bates Communication Inventory (MCDI)
* Unified Parkinson's Disease Rating Scale (UPDRS)
* Quick Neurological Screening Test 2nd Edition (QNST-2)
* Gait Analysis with motion capture video systems and interactive 3-dimensional modeling systems

ELIGIBILITY:
Inclusion Criteria:

* 5 to 12 years old
* pathogenic deletions or mutations of the SHANK3 gene
* stable medication regimens for at least three months prior to enrollment

Exclusion Criteria:

* closed epiphyses
* active or suspected neoplasia
* intracranial hypertension
* hepatic insufficiency
* renal insufficiency
* cardiomegaly / valvulopathy
* history of allergy to IGF-1 or any component of the formulation (mecasermin)
* history of extreme prematurity (<1000 grams) with associated early neo-natal complications, e.g. intra-cerebral hemorrhage, prolonged hypoxia, prolonged hypoglycemia
* patients with comorbid conditions deemed too medically compromised to tolerate the risk of experimental treatment with IGF-1

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2012-02; Primary Completion 2016-08-23 (Actual); Study Completion 2016-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kolevzon, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Seaver Austin Center, Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Kolevzon A, Bush L, Wang AT, Halpern D, Frank Y, Grodberg D, Rapaport R, Tavassoli T, Chaplin W, Soorya L, Buxbaum JD. A pilot controlled trial of insulin-like growth factor-1 in children with Phelan-McDermid syndrome. Mol Autism. 2014 Dec 12;5(1):54. doi: 10.1186/2040-2392-5-54. eCollection 2014. PMID 25685306
- [Derived] Kolevzon A, Breen MS, Siper PM, Halpern D, Frank Y, Rieger H, Weismann J, Trelles MP, Lerman B, Rapaport R, Buxbaum JD. Clinical trial of insulin-like growth factor-1 in Phelan-McDermid syndrome. Mol Autism. 2022 Apr 8;13(1):17. doi: 10.1186/s13229-022-00493-7. PMID 35395866
- See also: SHANK3 gene — http://www.shank3gene.org
- See also: Phelan-McDermid Syndrome Foundation — https://pmsf.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Study 1: Insulin-Like Growth Factor-1 (IGF-1) Then Normal Saline; Study 2: Insulin-Like Growth Factor-1 (IGF-1) Then Normal Saline: Insulin-Like Growth Factor-1 (IGF-1) and then placebo administered for 3 months with a four-week washout period in between. IGF-1 will be administered for 3 months subcutaneously.
- Study 1: Normal Saline Then IGF-1; Study 2: Normal Saline Then IGF-1: 12 weeks in each treatment arm (placebo and then IGF-1), separated by a 4-week wash-out phase
Period: Period 1: 12 Weeks
Arm/Group | Study 1: Insulin-Like Growth Factor-1 (IGF-1) Then Normal Saline | Study 1: Normal Saline Then IGF-1 | Study 2: Insulin-Like Growth Factor-1 (IGF-1) Then Normal Saline | Study 2: Normal Saline Then IGF-1
Started | 5 | 4 | 5 | 5
Completed | 5 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Washout 4 Weeks
Arm/Group | Study 1: Insulin-Like Growth Factor-1 (IGF-1) Then Normal Saline | Study 1: Normal Saline Then IGF-1 | Study 2: Insulin-Like Growth Factor-1 (IGF-1) Then Normal Saline | Study 2: Normal Saline Then IGF-1
Started | 5 | 4 | 5 | 5
Completed | 5 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Period 2: 12 Weeks
Arm/Group | Study 1: Insulin-Like Growth Factor-1 (IGF-1) Then Normal Saline | Study 1: Normal Saline Then IGF-1 | Study 2: Insulin-Like Growth Factor-1 (IGF-1) Then Normal Saline | Study 2: Normal Saline Then IGF-1
Started | 5 | 4 | 5 | 5
Completed | 5 | 3 | 5 | 5
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study 2: Insulin-Like Growth Factor-1 (IGF-1) Then Normal Saline: Participants who have pathogenic deletions or sequence variants of the SHANK3 gene.
  Insulin-Like Growth Factor-1 (IGF-1) and then placebo administered for 3 months with a four-week washout period in between. IGF-1 will be administered for 3 months subcutaneously.
- Total: Total of all reporting groups
Arm/Group | Study 1: Insulin-Like Growth Factor-1 (IGF-1) Then Normal Saline | Study 1: Normal Saline Then IGF-1 | Study 2: Insulin-Like Growth Factor-1 (IGF-1) Then Normal Saline | Study 2: Normal Saline Then IGF-1 | Total
Number analyzed (Participants) | 5 | 4 | 5 | 5 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.80 (4.64) | 6.90 (1.51) | 5.93 (1.06) | 6.97 (1.71) | 7.43 (2.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 1 | 10
  Male | 1 | 2 | 2 | 4 | 9
ABC-SW subscale score [Mean (Standard Deviation); unit: units on a scale] — 16 items on ABC-SW subscale, Each item is scored as 0 (never a problem), 1 (slight problem), 2 (moderately serious problem), or 3 (severe problem). Total score from 0 to 48 with higher score indicating poorer health outcomes.
  units on a scale | 20.4 (8.38) | 12.5 (7.72) | 19.2 (3.63) | 21 (6.36) | 18.58 (6.95)
Repetitive Behavior Scale (RBS) - Total [Mean (Standard Deviation); unit: units on a scale] — Total Score 43 items, each item scored on 4-point scale: 0-3, with total score from 0 (mild) to 129 (severe).
  The subscales are stereotyped behaviors 6 items (subscale 0-18), self-injurious behaviors 8 items (subscale 0-24), Compulsive behaviors- 8 items (subscale 0-24), Ritualistic Behaviors 6 items (subscale from 0-18), Sameness 11 items (subscale 0-33), restricted behaviors 4 items (subscale 0-12). Total score is the sum of all items in the subscale with total score range from 0 to 129. Higher scores indicate greater symptom severity.
  units on a scale | 35.4 (29.63) | 28 (16.10) | 12.4 (15.88) | 18 (9.92) | 23.21 (20.07)
Vineland Adaptive Behavior Composite Standard Score [Mean (Standard Deviation); unit: units on a scale] — Standardized scores on the Adaptive behavior composite range from 20-160 with higher scores indicating better functioning.
  units on a scale | 43.6 (13.67) | 47.75 (3.59) | 48.8 (5.81) | 49.2 (13.33) | 47.32 (9.80)

OUTCOME MEASURES:

1. Primary Outcome: Change in Aberrant Behavior Checklist - Social Withdrawal (ABC-SW) Subscale - Study 1
Description: 16 items on ABC-SW subscale, Each item is scored as 0 (never a problem), 1 (slight problem), 2 (moderately serious problem), or 3 (severe problem). Total score from 0 to 48 with higher score indicating poorer health outcomes.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Study 1: Insulin-Like Growth Factor-1 (IGF-1): IGF-1 (Increlex; Ipsen Biopharmaceuticals, Inc) is an aqueous solution for injection containing human insulin-like growth factor-1 (rhIGF-1) produced by recombinant DNA technology. Dose titration was initiated at 0.04 mg/kg twice daily by subcutaneous injection, and increased, as tolerated, every week by 0.04 mg/kg per dose to a maximum of 0.12 mg/kg twice daily.
- Study 1: Normal Saline: Placebo consisted of saline prepared in identical bottles by the research pharmacy at Mount Sinai.
Arm/Group | Study 1: Insulin-Like Growth Factor-1 (IGF-1) | Study 1: Normal Saline
Number analyzed (Participants) | 9 | 9
score on a scale
  Baseline | 15.78 (9.16) | 11.22 (7.29)
  Week 12 | 7.61 (5.71) | 9.70 (8.07)

2. Primary Outcome: Change in Aberrant Behavior Checklist - Social Withdrawal (ABC-SW) Subscale Study 2
Description: as for outcome 1
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Study 2: IGF-1: IGF-1 is an aqueous solution for injection containing human insulin-like growth factor-1 (Increlex; Ipsen Biopharmaceuticals, Inc)) produced by recombinant DNA technology. Dose titration was initiated at 0.04 mg/kg twice daily by subcutaneous injection, and increased, as tolerated, every week by 0.04 mg/kg per dose to a maximum of 0.12 mg/kg twice daily. Medication was administered subcutaneously twice daily with meals and glucose monitoring was performed by parents prior to each injection and at bedtime.
- Study 2: Placebo: Placebo consisted of saline prepared in identical bottles by the research pharmacy at Mount Sinai.
Arm/Group | Study 2: IGF-1 | Study 2: Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | -5.5 (7.46) | -6.3 (5.38)

3. Secondary Outcome: Change in Repetitive Behavior Scale - Study 2
Description: Repetitive Behavior Scale (RBS) - Total Score 43 items, each item scored on 4-point scale: 0-Behavior does not occur, 1-Behavior occurs and is a mild problem, 2-Behavior occurs and is a moderate problem, 3-Behavior occurs and is a severe problem. with total score from 0 (mild) to 129 (severe).
  The subscales are stereotyped behaviors 6 items (subscale 0-18), self-injurious behaviors 8 items (subscale 0-24), Compulsive behaviors- 8 items (subscale 0-24), Ritualistic Behaviors 6 items (subscale from 0-18), Sameness 11 items (subscale 0-33), restricted behaviors 4 items (subscale 0-12). Total score is the sum of all items in the subscale with total score range from 0 to 129. Higher scores indicate greater symptom severity.
Time Frame: Baseline and Week 12
Population: Participants in Study 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study 2: IGF-1 | Study 2: Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  RBS-Stereotyped Behavior | -0.3 (2.63) | -0.8 (2.19)
  RBS-Self-Injurious Behavior | -0.3 (1.64) | 0.2 (1.14)
  RBS-Compulsive Behavior | -0.8 (1.4) | 0.1 (0.88)
  RBS-Sameness Behavior | -1.4 (2.27) | -0.37 (1.74)
  RBS-Restricted Behavior | -1.1 (1.66) | -0.1 (1.29)
  RBS-Total | -3.5 (6.2) | -0.77 (5.73)

4. Secondary Outcome: Change in CGI-Improvement and Severity Scales; - Study 2
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study 2: IGF-1 | Study 2: Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  CGI - Severity | -0.2 (0.42) | -0.1 (0.32)
  CGI - Improvement | 2.6 (0.84) | 3.1 (1.28)

5. Secondary Outcome: Change in Caregiver Strain Questionnaire
Description: 21 question tool, about caregiver strain, where each question uses a Likert scale where 1 is "Not at all" and 5 is "Very much." The full scale ranges from 21-105, where higher scores indicate more severe strain.
Time Frame: Baseline and Week 12
Population: 4 participants missing data from at least one data point
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Study 2: Insulin-Like Growth: IGF-1 is an aqueous solution for injection containing human insulin-like growth factor-1 (Increlex; Ipsen Biopharmaceuticals, Inc)) produced by recombinant DNA technology. Dose titration was initiated at 0.04 mg/kg twice daily by subcutaneous injection, and increased, as tolerated, every week by 0.04 mg/kg per dose to a maximum of 0.12 mg/kg twice daily. Medication was administered subcutaneously twice daily with meals and glucose monitoring was performed by parents prior to each injection and at bedtime.
- Study 2: Normal Saline: Placebo consisted of saline prepared in identical bottles by the research pharmacy at Mount Sinai.
Arm/Group | Study 1: Insulin-Like Growth Factor-1 (IGF-1) | Study 1: Normal Saline | Study 2: Insulin-Like Growth | Study 2: Normal Saline
Number analyzed (Participants) | 9 | 9 | 6 | 10
score on a scale
  Baseline | 64.11 (17.32) | 63.22 (20.48) | 58 (18.89) | 55.00 (19.54)
  Week 12 | 61.11 (17.60) | 64.11 (17.08) | 55.67 (18.99) | 53.00 (19.68)

6. Secondary Outcome: Change in Sensory Profile (SP) - Study 2
Description: The SP is a standardized parent-completed questionnaire that assesses sensory processing and its impact on the functioning of children ages 3-10 yr. The 125 items represent behaviors that can be interpreted as responses to sensory experiences. The parent rates the observed frequency of these behaviors on a 5-point Likert scale (ranging from 1 always to 5 never). The tool consists of 14 sections, listed below, that refer to sensory processing, modulation, and behavioral and emotional responses. Subscale scores are listed below.
  Each section's raw score is compared with a threshold value to determine a category of performance: typical performance, probable difference (1 standard deviation below the mean), and definite difference (2 standard deviations below the mean). A lower raw score means a greater difference.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study 2: IGF-1 | Study 2: Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  SP-Auditory Processing (subscale range 8-40) | 1.6 (2.46) | 0.2 (2.39)
  SP-Visual Processing (subscale range 9-45) | 1.3 (4.92) | 1.5 (3.69)
  SP-Vestibular Processing (subscale range 11-55) | 0.9 (5.2) | -0.53 (4.06)
  SP-Touch Processing (subscale range 18-90) | 3.9 (4.89) | 0.3 (5.36)
  SP-Multisensory Processing (subscale range 7-35) | 0.9 (4.23) | -0.7 (3.68)
  SP-Oral Sensory Processing (subscale range 12-60) | 1 (5.08) | 0.5 (5.32)
  SP-Sensory Processing Related to Endurance/Tone (subscale range 9-45) | 0.5 (5.93) | 2 (3.33)
  SP-Modulation Related to Body Position and Movement (subscale range 10-50) | 5 (4.08) | -0.4 (3.24)
  SP-Modulation of Movement Affecting Activity Level (subscale range 7-35) | 0.2 (3.16) | 1.7 (5.58)
  SP-Modulation of Sensory Input Affecting Emotional Responses (subscale range 4-20) | -0.4 (1.17) | 0.6 (1.84)
  SP-Modulation of Visual Input Affecting Emotional Responses & Activity Level (subscale range 4-20) | 0.4 (1.65) | 0.9 (1.52)
  SP-Emotional/Social Responses (subscale range 17-85) | 3 (7.85) | 0.1 (5.3)
  SP-Behavioral Outcomes of Sensory Processing (subscale range 6-30) | 2.83 (6.59) | 0.11 (3.55)
  SP-Items Indicating Thresholds for Response (subscale range 3-15) | 1 (1.55) | 0 (2)

7. Secondary Outcome: Change in Short Sensory Profile (SSP) - Study 2
Description: The Short Sensory Profile is a caregiver report measure consisting of 38 items, each scored on a 1-point (always) to 5-point (never) Likert scale.
  SSP Subscales Tactile Sensitivity (7 to 35) Taste/Smell Sensitivity (4 to 20), Movement Sensitivity (3 to 15), Under-Responsive/Seek Sensation (7 to 35) , Auditory Filtering (6 to 30), Low Energy/Weak (6 to 30), Visual/Auditory Sensitivity (5 to 25), with total scale from (38 to 190)
  Lower scores indicate more sensory alterations.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study 2: IGF-1 | Study 2: Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  SSP-Tactile Sensitivity | 0.9 (2.73) | 0.7 (2.45)
  SSP-Taste/Smell Sensitivity | -0.2 (2.57) | -0.5 (1.08)
  SSP-Movement Sensitivity | 0.4 (1.26) | -0.3 (1.57)
  SSP-Underresponsive/Seeks Sensation | 2.87 (4.47) | -1.23 (3.61)
  SSP-Auditory Filtering | 0.9 (2.23) | 0.3 (2.67)
  SSP-Low Energy/Weak | -0.6 (3.89) | 1.36 (1.99)
  SSP-Visual/Auditory Sensitivity | 0.8 (1.23) | 0.8 (1.55)
  SSP-Total | 5.07 (11.43) | 1.13 (10.32)

ADVERSE EVENTS:
Time Frame: 28 weeks
Groups:
- Insulin-Like Growth Factor-1 (IGF-1): IGF-1 is an aqueous solution for injection containing human insulin-like growth factor-1 (Increlex; Ipsen Biopharmaceuticals, Inc)) produced by recombinant DNA technology. Dose titration was initiated at 0.04 mg/kg twice daily by subcutaneous injection, and increased, as tolerated, every week by 0.04 mg/kg per dose to a maximum of 0.12 mg/kg twice daily. Medication was administered subcutaneously twice daily with meals and glucose monitoring was performed by parents prior to each injection and at bedtime.
- Normal Saline: Placebo
Arm/Group | Insulin-Like Growth Factor-1 (IGF-1) | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 19/19 | 19/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin-Like Growth Factor-1 (IGF-1) (N=19) | Normal Saline (N=19)
Constipation (Gastrointestinal disorders) | 7 | 4
Sedation (Nervous system disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 5
Periobital/facial swelling (Skin and subcutaneous tissue disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 5
URTI (Infections and infestations) | 9 | 10
Sleep Disturbance (Nervous system disorders) | 11 | 7
Increased appetite (Metabolism and nutrition disorders) | 9 | 1
Mood changes/irritability (Nervous system disorders) | 9 | 8
Increased thirst (Metabolism and nutrition disorders) | 1 | 1
Increased phlegm (Infections and infestations) | 1 | 0
Teeth grinding (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Hand flapping (Nervous system disorders) | 1 | 0
Increased bowel movements (Gastrointestinal disorders) | 1 | 0
Increased chewing/biting (Nervous system disorders) | 2 | 0
Decreased visual acuity (Eye disorders) | 1 | 0
Lethargy/decreased energy (Nervous system disorders) | 6 | 4
Cooler body temperature/sweating (Nervous system disorders) | 1 | 0
Runny nose/congestion (Infections and infestations) | 7 | 8
Gait changes/fell (Nervous system disorders) | 3 | 5
Stomach virus (Infections and infestations) | 3 | 1
Anxiety (Nervous system disorders) | 0 | 2
Increased urine frequency (Renal and urinary disorders) | 2 | 0
Fever (Infections and infestations) | 7 | 5
Increased energy (Nervous system disorders) | 2 | 1
Gagging (Gastrointestinal disorders) | 2 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Erythema/swollen eyes (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Facial swelling (Skin and subcutaneous tissue disorders) | 2 | 0
Warmer body temperature (Endocrine disorders) | 2 | 1
Hair loss (Skin and subcutaneous tissue disorders) | 1 | 0
Increased aggression (Nervous system disorders) | 1 | 1
Hypoglycemia (Endocrine disorders) | 11 | 12
Stomach aches (Gastrointestinal disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Bruising at injection site (Skin and subcutaneous tissue disorders) | 1 | 0
Breast buds developed (Reproductive system and breast disorders) | 1 | 0
Bloody nose (Blood and lymphatic system disorders) | 1 | 2
Elevated heart rate (Cardiac disorders) | 0 | 1
Increased ear wax (Ear and labyrinth disorders) | 0 | 1
Increased reflux (Gastrointestinal disorders) | 1 | 1
Ear Infections (Infections and infestations) | 1 | 1
Broken bone (Injury, poisoning and procedural complications) | 0 | 1
Increased drooling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Increased eye rolling (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Redness around perineum (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The small sample size and expectancy bias due to relying on parent reported outcome measures may contribute to limitations in interpreting results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-01-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT01525901/Prot_SAP_000.pdf